CLINICAL TRIAL: NCT04933409
Title: 3D Printed Donor Tooth Replica in Autotransplantation of Teeth. A Randomized Clinical Trial.
Brief Title: 3D Printed Donor Tooth Replica in Autotransplantation of Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: College of Medical Sciences Teaching Hospital. Nepal (Other)
Responsible Party: Principal Investigator, Ashutosh Kumar Singh, Assistant Professor, College of Medical Sciences Teaching Hospital. Nepal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOM1
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Decayed Teeth
Keywords: decayed teeth; autotransplantation; 3d printing
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled tria
Who Masked: Outcomes Assessor
Masking Description: The outcomes will be evaluated by a blinded researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed replica of Donor tooth (Experimental): 3D printed replica of Donor tooth
  Interventions: Procedure: 3D printed replica of the donor tooth
- Conventional (Active Comparator): Conventional method of autotransplantation.
  Interventions: Procedure: Conventional Autotransplantation of tooth

INTERVENTIONS:
Procedure: 3D printed replica of the donor tooth — 3D printed replica of the donor tooth.
  Arms: 3D printed replica of Donor tooth
Procedure: Conventional Autotransplantation of tooth — Conventional Autotransplantation of tooth without using the 3D printed guide
  Arms: Conventional

SUMMARY:
3D printed replicas of the donor tooth can reduce extraoral time during the autotransplantation of teeth, which can reduce dehydration and manipulation of periodontal tissue of the donor tooth, thus possibly increasing the success rate.

DETAILED DESCRIPTION:
This technique of autotransplantation has been innovated using 3-dimensional (3D) imaging and rapid prototyping.The use of a 3D-printed replica of the donor tooth is thought to minimize the risk of iatrogenic damage to the actual donor tooth. Nevertheless, no large prospective and comparative studies are available to assess the outcomes using these 3D techniques. Therefore, this study aimed to compare 3D printed replicas in autotransplantation of teeth, compared to the conventional technique. The present study will evaluate the feasibility, clinical satisfied accuracy, and stability of a novel approach for computer-aided autotransplantation of teeth. This new approach facilitated the surgical procedure and might be a viable and predictable method for autotransplantation of teeth.

Application of printed 3D replicas of transplanted teeth facilitates surgical preparation of the recipient site, shortens the extra-alveolar time, and reduces the minimum the number of attempts of the donor tooth insertion at the prepared socket. Their use can significantly decrease the risk of damage to the root surface of a transplant, thus increasing the chance of success.

ELIGIBILITY:
Inclusion Criteria:

1. patient presenting with decayed first molars
2. autotransplantation of third molar at the recipient site

Exclusion Criteria:

1. Diabetic, pregnant patients
2. other autotransplantations (other than first molar recipient and third molar donor)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of teeth that fail | two weeks
  reduced mobility (less than grade II) after 2 weeks of autotransplantation
Operative time | 1 day
  Operative time from the start of socket preparation at the recipient site
Rate of Ankylosis (replacement resorption) | 6 months
  Ankylosis (replacement resorption)
Rate of root resorption | 6 months
  infection related root resorption

SECONDARY OUTCOMES:
Cost difference of the treatment | 1 day
  Cost of 3D printing

IPD SHARING:
Plan to Share IPD: Yes
Yes, On request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year
Access Criteria: On request to the principal investigator